CLINICAL TRIAL: NCT05011227
Title: A Prospective, Single-arm, Multi-center Clinical Study of Camrelizumab and Chemotherapy Combined With Endoscopic Surgery in the Treatment of Recurrent Nasopharyngeal Carcinoma
Brief Title: Camrelizumab and Chemotherapy Combined With Endoscopic Surgery for Recurrent Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rNPC-SA-Neo-Cam-V1
Record Dates: First submitted 2021-08-07; First posted 2021-08-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: endoscopic surgery; Inductive chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Drug Therapy; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab and chemotherapy combined with endoscopic surgery (Experimental): Camrelizumab and chemotherapy combined with endoscopic surgery
  Interventions: Drug: Camrelizumab; Drug: Chemotherapy; Procedure: endoscopic surgery

INTERVENTIONS:
Drug: Camrelizumab — 2 cycles Camrelizumab before endoscopic surgery and one year after
Drug: Chemotherapy — 2 cycles Gemcitabine based chemotherapy before endoscopic surgery, with or without after surgery
Procedure: endoscopic surgery — standard endoscopic surgery for recurrent nasopharyngeal carcinoma

SUMMARY:
To explore the effect of Camrelizumab and chemotherapy combining with endoscopic surgery in the treatment of recurrent nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed recurrent nasopharyngeal carcinoma
* American Joint Committee on Cancer recurrent rT2(recurrent T2)(including deep parapharyngeal space), recurrent T3, recurrent T4 which can be surgically removed
* Age ≥18 years old
* Informed consent signed
* With or without lymph node metastasis, which can be surgically removed
* No massive hemorrhage risk recently
* No distant metastasis
* ≥6 months from initial radiotherapy to recurrence
* Radical radiation only once
* Sufficient organ function
* Eastern Cooperative Oncology Group score 0-2

Exclusion Criteria:

* With a history of allergic to platinum drugs and similar compounds
* Evidence of distant metastasis or radiation encephalopathy or leptomeningeal disease (LMD)
* Have received radioactive seed implantation in the treatment area
* Suffer from uncontrolled disease which could interfere with treatment
* Suffered from another malignant tumor or multiple primary tumors at the same time within 5 years (excluding fully treated basal cell or squamous cell skin cancer, cervical cancer in situ, etc.)
* The patient has surgical contraindications: such as severe cardiopulmonary disease, coagulation dysfunction and so on
* The patients have autoimmune diseases
* The patient is using immunosuppressive agents or systemic glucocorticoid to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other), and continues to use it within 2 weeks before the first administration
* Severe allergic reaction to other monoclonal antibodies
* Previously received PD-1 monoclonal antibody, CTLA-4 monoclonal antibody (or any other antibody that acts on T cell co-stimulation or checkpoint pathway) treatment
* Live vaccines have been inoculated within 4 weeks before the first administration or during the study period
* The patient has any situation that may hinder study compliance or the safety during the study period
* Existence of serious neurological or psychiatric diseases, such as dementia and seizures
* Uncontrolled active infection
* Pregnant or breastfeeding women
* Those who have no personal freedom and independent capacity for civil conduct
* There are other situations that are not suitable for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of first treatment until the date of death from any cause, up to 4 years.
  2 year Overall Survival rate

SECONDARY OUTCOMES:
Local recurrence free survival | From date of first treatment until the date of local recurrence or death from any cause, up to 4 years.
  the date of first treatment to local failure or death
Progression free survival | From date of first treatment until the date of disease progression or death from any cause, up to 4 years.
  the date of first treatment to the first recording of disease progression or death from any cause.
Rate of negative margin | At the time of pathology reporting, util the pathology report of last subject was completed, up to 2.5 years.
  negative margin rate according to pathology report
distant metastasis free survival | From date of first treatment until the date of distant metastasis or death from any cause, up to 4 years.
  the date of first treatment to distant metastasis or death
pathologic complete remission | At the time of pathology reporting,util the pathology report of last subject was completed, up to 2.5 years.
  pathologic complete remission

OTHER OUTCOMES:
quality of life-（EORTC QLQ) - C30 version3.0 | From date of first treatment to the end of study, at each visit, up to 4 years.
  using European Organisation for Research and Treatment of Cancer quality of life questionaire（EORTC QLQ) - C30 version3.0. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
quality of life-（EORTC QLQ) - H&N35 | From date of first treatment to the end of study, at each visit, up to 4 years.
  using European Organisation for Research and Treatment of Cancer quality of life questionaire（EORTC QLQ）- H&N35，All of the scales and single-item measures range in score from 0 to 100. For all the scales and single-items a high score represents a high level of symptomatology or problems.
adverse effect | From date of first treatment to the end of study, up to 4 years.
  Using CTCAE Version5.0 to evaluate related adverse effect
immune related adverse effect | From date of first treatment to the end of study, up to 4 years.
  Using CTCAE Version5.0 to evaluate immune related adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD,PHD, Principal Investigator — Eye&ENT Hospital,Fudan University
Locations (7):
- China (7):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Eye& ENT Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR